CLINICAL TRIAL: NCT06872086
Title: Assessment of Blood Indices As Predictors of Disease Activity in Systemic Lupus Erythematosus
Brief Title: Assessment of Blood Indices in Systemic Lupus Erythematosus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Ibrahim Altayeb Sayed, resident at the internal medicine department, Assiut University
Other Study IDs: blood indices in SLE
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: SLE; Blood Indices
Keywords: SLE; Systemic Lupus Erythematosus; Blood Indices
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SLE Patients: This group consists of 70 adult patients diagnosed with systemic lupus erythematosus (SLE) according to the 2019 ACR/EULAR classification criteria. These participants will undergo clinical assessments to evaluate disease activity using the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K). Blood indices, including lymphocyte-monocyte ratio (LMR), neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), and systemic immune-inflammatory index (SIRI), will be analyzed to investigate their correlation with disease activity.
- Healthy Controls: This group includes 70 age- and gender-matched healthy individuals without autoimmune diseases or significant comorbidities. Participants will serve as controls for comparison of blood indices, including LMR, NLR, PLR, and SIRI, to establish baseline values and assess differences between healthy individuals and SLE patients.

SUMMARY:
This case-control study aims to explore the relationship between specific blood indices (lymphocyte-monocyte ratio, neutrophil-to-lymphocyte ratio, platelet-to-lymphocyte ratio, and systemic immune-inflammatory index) and disease activity in patients with systemic lupus erythematosus (SLE).

The study includes 70 SLE patients and 70 healthy controls, matched for age and gender, recruited from Assiut University Hospital.

Disease activity is assessed using the SLEDAI-2K score, and blood indices are analyzed to determine correlations with disease activity.

DETAILED DESCRIPTION:
This case-control study will be conducted at Assiut University Hospital, involving 70 patients diagnosed with SLE according to the 2019 ACR/EULAR classification criteria and 70 healthy controls matched for age and gender. Inclusion criteria include patients aged 18 years or older with SLE, while exclusion criteria include other autoimmune diseases, recent infections, and hematological disorders unrelated to SLE.

Study Tools and Procedures:

Demographic Information: Collect data on age, gender, duration of illness, and relevant medical history.

Clinical Assessment: Disease activity will be evaluated using the SLEDAI-2K score, which includes parameters such as mucocutaneous manifestations, musculoskeletal symptoms, renal involvement, neurological symptoms, and hematological abnormalities.

Laboratory Tests: A complete blood count (CBC) will be performed to obtain lymphocyte, monocyte, neutrophil, and platelet counts. Additional tests may include serum creatinine levels, urinalysis for proteinuria, 24-hour urinary proteins, CRP, ESR, and complement levels (C3, C4) to assess overall disease status.

Study Tools: The SLEDAI-2K tool will categorize patients based on their disease activity levels. CBC results will be analyzed to calculate LMR, NLR, PLR, and SIRI, which will be correlated with the SLEDAI-2K score.

Research Outcome Measures Primary Outcome: The primary objective is to assess the correlation between blood indices (LMR, NLR, PLR, SIRI) and SLE disease activity as measured by the SLEDAI-2K score. This will involve statistical analysis to determine if there is a significant correlation between these indices and disease activity.

Secondary Outcomes:

Comparison of Blood Indices: Evaluate differences in LMR, NLR, PLR, and SIRI between SLE patients and healthy controls.

Disease Activity Variability: Analyze how variations in blood indices correlate with changes in SLEDAI-2K scores over time.

Exploration of Additional Hematological Indices: Investigate other hematological parameters such as mean platelet volume (MPV) to determine their association with disease activity.

Impact of Treatment: Assess how treatment interventions affect blood indices and correlate these changes with improvements or deteriorations in SLEDAI-2K scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older diagnosed with SLE according to the 2019 ACR/EULAR classification criteria.
* Healthy controls without any autoimmune diseases or significant comorbidities

Exclusion Criteria:

* • Patients with other autoimmune diseases (e.g., rheumatoid arthritis, Sjögren's syndrome).

  * Recent infections or acute inflammatory conditions.
  * Individuals with hematological disorders unrelated to SLE (e.g., leukemia, lymphoma).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cases are Patients aged 18 years or older diagnosed with SLE according to the 2019 ACR/EULAR classification criteria and • Healthy controls without any autoimmune diseases or significant comorbidities
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between Blood Indices and SLEDAI -2K score | 1 month
  The primary outcome of this study will be to assess the relationship between lymphocyte-monocyte ratios (LMR), neutrophil-to-lymphocyte ratios (NLR), platelet-to-lymphocyte ratios (PLR), systemic immune-inflammatory index (SIRI) and systemic lupus erythematosus disease activity as measured by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K). This will involve statistical analysis to determine if there is a significant correlation between these blood indices and the SLEDAI-2K score, indicating their potential utility as biomarkers for SLE activity.

IPD SHARING:
Plan to Share IPD: No